CLINICAL TRIAL: NCT05853081
Title: Prognostic Value of the Fat-free Mass Index on a Multidimensional Scale in Chronic Obstructive Pulmonary Disease
Brief Title: FODEPOC Study: Fat-free Mass Index in Copd
Acronym: FODEPOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Daniel López Padilla, Clinical Professor Daniel López Padilla, Hospital General Universitario Gregorio Marañon
Other Study IDs: FODEPOC
Record Dates: First submitted 2023-03-02; First posted 2023-05-10 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; prognosis; nutrition assessment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FEV1 < 30%: open groups with forced expiratory flow in the first second (FEV1) < 30%. It will be followed for at least two years.The fat-free mass index (FFMI) will be measured instead of the body mass index (BMI) with bioelectrical impedance analysis.
  Interventions: Diagnostic Test: Bioelectrical impedance analysis
- FEV1 30-50%: open groups with forced expiratory flow in the first second (FEV1) < 30%. It will be followed for at least two years.The fat-free mass index (FFMI) will be measured instead of the body mass index (BMI) with bioelectrical impedance analysis.
  Interventions: Diagnostic Test: Bioelectrical impedance analysis
- FEV1 > 50%: open groups with forced expiratory flow in the first second (FEV1) < 30%. It will be followed for at least two years.The fat-free mass index (FFMI) will be measured instead of the body mass index (BMI) with bioelectrical impedance analysis.
  Interventions: Diagnostic Test: Bioelectrical impedance analysis

INTERVENTIONS:
Diagnostic Test: Bioelectrical impedance analysis — The Fat-free mass index (FFMI) will be measured using bioelectrical impedance analysis. Exacerbations and mortality will be recorded during follow-up to evaluate the prognostic value of the FODE scale.

SUMMARY:
General Objective: To compare the prognostic value of the FODE scale for COPD exacerbations, where the fat-free mass index (FFMI) will be measured instead of the body mass index (BMI) in the BODE scale. Specific objectives: to describe the nutritional status of COPD patients according by the GesEPOC and GOLD phenotypes; to compare the mortality prognostic value of FODE with BODE; to compare the exacerbations and mortality prognostic value of the BODCAT scale, which includes the CAT questionnaire instead of the six-minute walking test (6MWT), with BODE; to compare the mortality prognostic value of the FODE and FODEx scales, where the BMI and the 6MWT will be substituted by the FFMI and the severe exacerbations in the previous year, respectively, with BODE and BODEx. Methods: prospective, with no intervention besides the recommendations of COPD clinical guidelines, where patients will be allocated into three parallel and open groups according to their forced expiratory flow in the first second (FEV1) in the fashion FEV1 < 30%: FEV1 30-50% : FEV1 > 50%, and will be followed for at least two years. FFMI will be measured using bioelectrical impedance analysis. Exacerbations and mortality will be recorded during follow-up to evaluate the prognostic value of the FODE scale, which hypothetically will increase in 10% the prognostic value of the BODE scale.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Chronic obstructive pulmonary disease (COPD) is a respiratory disease characterized by chronic airflow limitation with significant systemic effects, which is often associated with one or more comorbidities such as malnutrition with negative effects on the evolution of the disease and increased risk of mortality. To determine the prognostic severity of COPD, Celli et al. proposed in 2004 the BODE index, a multidimensional scale that integrates information on body mass index (BMI), forced expiratory volume in the first second (FEV1), dyspnea and exercise capacity, evaluated by the 6-minute walking test (6MWT). Except for BMI, to which it assigns a maximum value of 1 point, it assigns from 0 to 3 points in the rest of the items, so the highest possible score is 10. The BODE reflects the progressive modification of the disease and is useful for predicting hospitalization and the risk of death among patients with COPD, and an increase at one point is associated with an increase of 34% of all causes of mortality and 62% due to respiratory causes.

The BODE index uses BMI as a variable of the nutritional status of subjects with COPD, however, alterations in body composition may occur, in the absence of clinically significant weight loss. In patients with COPD, a lower fat-free mass index (FFMI) contributes to worsening lung function, quality of life and exercise capacity, as well as a negative impact on exacerbations and survival, suggesting that FFMI may be more accurate than BMI as a prognostic factor for mortality in these patients. In a recent study conducted by Luo Y et al., the nutritional status of patients with stable COPD was evaluated, showing that 48.5% patients had a low FFMI (≤15 kg/m2 in women and ≤16 kg/m2 in men) with a significantly greater decrease in those with more advanced disease. The FFMI (Fat free mass index) can be objectively measured by electrical bioimpedance analysis (BIA), dual-energy X-ray absorptiometry, computed tomography, ultrasonography or magnetic resonance imaging. The BIA is based on the Relationship between the electrical properties of the human body, the body composition of the different tissues and the total water content in the body. It is a simple, cheap, easy to perform and non-invasive method, based on the resistance to the passage of electric current through the body compartments and very useful for performing body composition analysis.

On the other hand, the 6MWT is a predictor of mortality in patients with COPD. Although it is a widely used test that impresses to be simple, its forecasting reliability depends on strict repeatability conditions and qualified human resources which presents obvious difficulties in people with walking disabilities and elders. To facilitate the multidimensional approach to this disease, other simpler, adequately validated and accepted clinical tools have been developed to estimate the severity of symptoms and their impact on quality of life. The COPD Assessment test (CAT) is the most widely used in clinical practice guidelines and is a questionnaire consisting of eight domains with a score of 1 to 5, which measure the health status of patients with COPD in such a way that the higher the score, the worse the patient's condition. According to the latest GOLD guide, it is an indispensable variable to classify the severity of the disease with a cut-off point in the 10 points. Its prognostic value has been widely demonstrated, and a recent study showed that patients with severe COPD and a CAT ≥ 15 have a significantly higher risk of exacerbations. Another multidimensional scale proposed in the literature is the BODEx, which also addresses the need to simplify the tests to be performed, considering the technical and administrative difficulties of the 6MWT, and proposed in 2009 by Soler-Cataluña et al., in which they found a prognostic mortality value similar to the BODE without the need to perform the 6MWT because it would be replaced by the number of serious exacerbations (those that required hospital care) in the previous year. Although the BODE index is widely used in clinical practice, it is believed that its performance can be improved. For example, with respect to its application as an indication for lung transplantation, the previous BODE has not demonstrated a prognostic value of the overall post-transplant results except in the subgroup of patients with a BODE ≥ 7. Therefore, with the hypothesis of being able to implement other items other than the scale, more representative in terms of nutritional status (FFMI instead of BMI) and simpler (the CAT instead of the 6MWT), the main objective is to compare the prognostic value of the multidimensional FODE scale (F of fat-free mass index), which replaces the BMI with the FFMI, compared to the BODE scale. As a secondary objective to analyse the variants in which the 6MWT is replaced by the CAT questionnaire.

STUDY HYPOTHESIS

* Conceptual Hypothesis On the multidimensional BODE scale, the Fat Free Mass Index is a better prognostic factor for exacerbations and mortality in COPD patients, compared to the Body Mass Index.
* Operational Hypothesis The Fat Free Mass Index better predicts exacerbations and mortality of COPD patients compared to the Body Mass Index, increasing by 10% of the area below the ROC curve of the multidimensional BODE scale.

METHODOLOGY

Population and sample size. The target population will be consecutive patients over 40 years of age with a history of tobacco use with a package-years index greater than or equal to 10. According to the latest epidemiological studies, the prevalence of COPD in the general population is around 12%, and based on the prevalence of malnutrition in this population, measured by the Fat Free Mass Index ranging between 4 and 35%, it is proposed from the following calculation of the sample for survival studies with a predictable correlation with other factors in a predictable Cox multivariate analysis: Relative risk to detect 1.5 Proportion of exposed subjects 0.48 Censored observations proportion 0 Confidence level 0.95 Statistical power 0.8 Other factors correlation to include in the model 0.28 Lost to follow-up percentage 0.15 Minimum sample size 237

Study design: Observational, prospective and multicentre study, which will determine in the cohort of patients with a recent diagnosis of COPD, the prognostic value of the nutritional parameter of Fat Free Mass Index (FFMI) on a multidimensional scale in which it will replace the Body Mass Index (BMI), and the parameters of Forced Exhaled Volume in the first second (FEV1) will be maintained, dyspnea as measured by the Modified Medical Research Council (mMRC) scale, and exercise capacity measured with the 6MWT. Like the BODE study5, a follow-up of the cohort of no less than two years is proposed with a periodicity of reviews between three and six months. Four groups will be proposed according to the quartiles of the FODE index obtained, following the methodology of the study proposed by the BODE index. The low FFMI cut-off point was set at 15 kg/m2 in women and 16 kg/m2 in men, used in previous studies9. On the other hand, the BODEx index will be calculated according to what was proposed by its creators, in which the item will have a score of 0 to 2 points as follows: no exacerbations = 0 points; 1 to 2 severe exacerbations in the last year = 1 point; and 3 or more exacerbations = 2 points16. To guarantee the representativeness of the severity of COPD, the inclusion of patients in the 1:1:1 sense is proposed with the following three groups: group with FEV1 greater than or equal to 50%, patients with FEV1 greater than or equal to 30% and less than 50%, and patients with an FEV1 less than 30%.

Bioelectrical impedance analysis (BIA). BIA is based on the relationship between the electrical properties of the human body, the body composition of different tissues and the total water content in the body. For FFMI calculation, the TANITA body composition monitor model® BC-545, a brand used in recent studies and a model specifically validated in the Spanish population, will be used as an adequate meter for body composition with an adequate agreement with other tetrapolar BIA monitors, specifically the BodyStat® 1500 model, used in other recent publications. Description of the technique: Body composition monitor scale, InnerScanSegmental, digital, TANITA Brand® BC-545, offers information on the percentage of total body fat and muscle mass by body segments: right arm, left arm, right leg, left leg and trunk, in addition to informing us about the basal metabolic rate, fat-free weight, bone weight (PO) and visceral fat. The BIA measures body composition by sending a low-frequency, safe signal throughout the body, from the base of the scale. This signal circulates freely among the fluid of the muscle tissue though encounters the resistance of the fatty tissue. This resistance, the bioimpedance, is measured accurately and its results are contrasted according to the sex, height, and weight of the person to calculate in a personalized way the fat reading and body composition. To take the measurement with the scale, the barefoot subject places the feet each on an electrode and makes use of the retractable cable system, which transmits a small electric current that runs through the body passing through all the body tissue more slowly through fat than through muscle.

Statistical analysis and measurements. Statistical analysis will be performed using SPSS version 21.0 (SPSS Inc., Chicago, IL). Qualitative variables will be presented as absolute numbers and percentages, while quantitative variables as means ± standard deviations, ranges, medians or interquartile ranges as the case may be. The normal distribution of the variables will be evaluated with the Kolmogorov-Smirnov test. The difference between the dichotomous characteristics will be analysed with the Chi-Square test with fisher's exact correction, and the quantitative variables by the ANOVA test in the case of reaching normality or the Kruskal-Wallis test when it is not achieved. The outcome variables will be death and exacerbations. The cumulative survival analysis will be performed using the Kaplan-Meier test and the comparative curves using the log-rank test. For the diagnostic validation of the FODE scale, Receiver Operating Characteristics (ROC) Curves will be used and compared with that of the BODE. The variables considered relevant according to similar previous studies, and the statistical significance presented in the univariate analysis previously described, will be analysed in a Cox proportional risk model to determine the independent association with mortality and exacerbations in the four groups formed. Finally, to verify the assumption of proportional risks, diagnostic and residual analyses will be carried out. As a sensitivity analysis, the prognostic value of the FODE scale will be analysed according to the phenotype and severity classifications of the latest GOLD and GesEPOC guidelines. In all analyses, statistical significance shall be set at a p-value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Man or woman > 40 years.
* Smoker or former smoker with a pack-years index ≥ 10.
* COPD diagnosis of at least 2 years prior to inclusion in the study, according to the following spirometry criteria: airflow obstruction documented by spirometry after bronchodilator treatment and in the clinical stability phase, with an forced expiratory volume in the first second / forced vital capacity (FEV1/FVC) ratio of less than 0.7, based on the latest GOLD and GesEPOC guidelines.1,14
* Clinical stability will always be defined according to the following criteria:
* No evidence of change in COPD maintenance treatment in the 4 weeks prior to inclusion in the study.
* No evidence of exacerbation that required the use of systemic antibiotics and/or corticosteroids in at least 4 weeks prior to inclusion in the study.
* Patients should be able to perform all procedures necessary for the study at the discretion of the investigator, including: acceptable and reproducible spirometry; 6-minute walking test; bioelectrical impedance analysis

Exclusion Criteria:

* Patients with another significant disease other than COPD (neoplastic, cardiovascular, metabolic, infectious or any clinical condition) as a foreseeable cause of death in the period of less than one year or that may cause a significant alteration of the nutritional status of the patient.
* Taking nutritional supplements and / or anabolic drugs in the last 12 months.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: population will be selected from pulmonology hospital consultations
Sampling Method: Probability Sample
Enrollment: 237 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fat Free Mass Index | Baseline
  Weight in kilograms and body fat percentage will be measured by bioelectrical impedance analysis, and height in meters. Weight, height and boday fat percentage will be combined to report Fat Free Mass Index.
Incidence of exacerbations | 12 months after inclusion
  Total frequency of exacerbations, frequency of exacerbations that required hospitalization and exacerbations free period since baseline.
Forced Expiratory Volumen in the first second | Baseline
  Mililiters of expired volume in the first second during a forced spirometry
Body Mass Index | Baseline
  Weight in kilograms and and height in meters. Weight and height will be combined to report Body Mass Index
Dyspnea | Baseline, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months after inclusion
  Dyspnea degree measured by the modified Medical Research Council Dyspnea Scale. Score ranges from 0 to 4, higher scores indicate worse dyspnea.
6 minute walking test | Baseline, 1 year, 2 years, 3 years
  Distance covered during 6 minutes of walking, measured in meters

SECONDARY OUTCOMES:
Changes in COPD clinical status | Baseline, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months after inclusion
  COPD Assesment Tool
Incidence of mortality | Baseline, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months after inclusion
  Total frequency of deaths, frequency of deaths due to respiratory cause and death free period since baseline.
COPD health related quality of life | Baseline, 1 year, 2 years, 3 years
  St. Georges´ Questionnaire to assess health related quality of life. Scores range from 0 to 100, with higher scores indicating more limitations
Major cardiovascular events | Baseline, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months after inclusion
  Frequency of stroke, acute myocardial infarction and heart failures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Not applicable since the study is not a clinical trial.

REFERENCES:
- [Background] Luo Y, Zhou L, Li Y, Guo S, Li X, Zheng J, Zhu Z, Chen Y, Huang Y, Chen R, Chen X. Fat-Free Mass Index for Evaluating the Nutritional Status and Disease Severity in COPD. Respir Care. 2016 May;61(5):680-8. doi: 10.4187/respcare.04358. Epub 2016 Jan 26. PMID 26814217
- [Result] Miravitlles M, Soler-Cataluna JJ, Calle M, Molina J, Almagro P, Quintano JA, Trigueros JA, Cosio BG, Casanova C, Antonio Riesco J, Simonet P, Rigau D, Soriano JB, Ancochea J. Spanish Guidelines for Management of Chronic Obstructive Pulmonary Disease (GesEPOC) 2017. Pharmacological Treatment of Stable Phase. Arch Bronconeumol. 2017 Jun;53(6):324-335. doi: 10.1016/j.arbres.2017.03.018. Epub 2017 May 3. English, Spanish. PMID 28477954
- [Result] Vanfleteren LE, Spruit MA, Groenen M, Gaffron S, van Empel VP, Bruijnzeel PL, Rutten EP, Op 't Roodt J, Wouters EF, Franssen FM. Clusters of comorbidities based on validated objective measurements and systemic inflammation in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Apr 1;187(7):728-35. doi: 10.1164/rccm.201209-1665OC. PMID 23392440
- [Result] Celli BR, Decramer M, Wedzicha JA, Wilson KC, Agusti A, Criner GJ, MacNee W, Make BJ, Rennard SI, Stockley RA, Vogelmeier C, Anzueto A, Au DH, Barnes PJ, Burgel PR, Calverley PM, Casanova C, Clini EM, Cooper CB, Coxson HO, Dusser DJ, Fabbri LM, Fahy B, Ferguson GT, Fisher A, Fletcher MJ, Hayot M, Hurst JR, Jones PW, Mahler DA, Maltais F, Mannino DM, Martinez FJ, Miravitlles M, Meek PM, Papi A, Rabe KF, Roche N, Sciurba FC, Sethi S, Siafakas N, Sin DD, Soriano JB, Stoller JK, Tashkin DP, Troosters T, Verleden GM, Verschakelen J, Vestbo J, Walsh JW, Washko GR, Wise RA, Wouters EF, ZuWallack RL; ATS/ERS Task Force for COPD Research. An Official American Thoracic Society/European Respiratory Society Statement: Research questions in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2015 Apr 1;191(7):e4-e27. doi: 10.1164/rccm.201501-0044ST. PMID 25830527
- [Result] Vestbo J, Prescott E, Almdal T, Dahl M, Nordestgaard BG, Andersen T, Sorensen TI, Lange P. Body mass, fat-free body mass, and prognosis in patients with chronic obstructive pulmonary disease from a random population sample: findings from the Copenhagen City Heart Study. Am J Respir Crit Care Med. 2006 Jan 1;173(1):79-83. doi: 10.1164/rccm.200506-969OC. PMID 16368793
- [Result] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Result] Schols AM, Ferreira IM, Franssen FM, Gosker HR, Janssens W, Muscaritoli M, Pison C, Rutten-van Molken M, Slinde F, Steiner MC, Tkacova R, Singh SJ. Nutritional assessment and therapy in COPD: a European Respiratory Society statement. Eur Respir J. 2014 Dec;44(6):1504-20. doi: 10.1183/09031936.00070914. Epub 2014 Sep 18. PMID 25234804
- [Result] de Blasio F, Di Gregorio A, de Blasio F, Bianco A, Bellofiore B, Scalfi L. Malnutrition and sarcopenia assessment in patients with chronic obstructive pulmonary disease according to international diagnostic criteria, and evaluation of raw BIA variables. Respir Med. 2018 Jan;134:1-5. doi: 10.1016/j.rmed.2017.11.006. Epub 2017 Nov 17. PMID 29413494
- [Result] de Blasio F, Scalfi L, Di Gregorio A, Alicante P, Bianco A, Tantucci C, Bellofiore B, de Blasio F. Raw Bioelectrical Impedance Analysis Variables Are Independent Predictors of Early All-Cause Mortality in Patients With COPD. Chest. 2019 Jun;155(6):1148-1157. doi: 10.1016/j.chest.2019.01.001. Epub 2019 Jan 17. PMID 30659818
- [Result] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486
- [Result] Lukaski HC, Bolonchuk WW, Hall CB, Siders WA. Validation of tetrapolar bioelectrical impedance method to assess human body composition. J Appl Physiol (1985). 1986 Apr;60(4):1327-32. doi: 10.1152/jappl.1986.60.4.1327. PMID 3700310
- [Result] Redelmeier DA, Bayoumi AM, Goldstein RS, Guyatt GH. Interpreting small differences in functional status: the Six Minute Walk test in chronic lung disease patients. Am J Respir Crit Care Med. 1997 Apr;155(4):1278-82. doi: 10.1164/ajrccm.155.4.9105067.
- [Result] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Result] Singh D, Agusti A, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Criner GJ, Frith P, Halpin DMG, Han M, Lopez Varela MV, Martinez F, Montes de Oca M, Papi A, Pavord ID, Roche N, Sin DD, Stockley R, Vestbo J, Wedzicha JA, Vogelmeier C. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease: the GOLD science committee report 2019. Eur Respir J. 2019 May 18;53(5):1900164. doi: 10.1183/13993003.00164-2019. Print 2019 May. PMID 30846476
- [Result] Jo YS, Yoon HI, Kim DK, Yoo CG, Lee CH. Comparison of COPD Assessment Test and Clinical COPD Questionnaire to predict the risk of exacerbation. Int J Chron Obstruct Pulmon Dis. 2017 Dec 22;13:101-107. doi: 10.2147/COPD.S149805. eCollection 2018. PMID 29317814
- [Result] Soler-Cataluna JJ, Martinez-Garcia MA, Sanchez LS, Tordera MP, Sanchez PR. Severe exacerbations and BODE index: two independent risk factors for death in male COPD patients. Respir Med. 2009 May;103(5):692-9. doi: 10.1016/j.rmed.2008.12.005. Epub 2009 Jan 7. PMID 19131231
- [Result] Lahzami S, Bridevaux PO, Soccal PM, Wellinger J, Robert JH, Ris HB, Aubert JD. Survival impact of lung transplantation for COPD. Eur Respir J. 2010 Jul;36(1):74-80. doi: 10.1183/09031936.00087809. Epub 2009 Dec 8. PMID 19996194
- [Result] Nyberg A, Saey D, Maltais F. Why and How Limb Muscle Mass and Function Should Be Measured in Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2015 Sep;12(9):1269-77. doi: 10.1513/AnnalsATS.201505-278PS. PMID 26208090
- [Result] Mete B, Pehlivan E, Gulbas G, Gunen H. Prevalence of malnutrition in COPD and its relationship with the parameters related to disease severity. Int J Chron Obstruct Pulmon Dis. 2018 Oct 11;13:3307-3312. doi: 10.2147/COPD.S179609. eCollection 2018. PMID 30349235
- [Result] McDonald MN, Diaz AA, Rutten E, Lutz SM, Harmouche R, San Jose Estepar R, Kinney G, Hokanson JE, Gower BA, Wouters EFM, Rennard SI, Hersh CP, Casaburi R, Dransfield MT, Silverman EK, Washko GR. Chest computed tomography-derived low fat-free mass index and mortality in COPD. Eur Respir J. 2017 Dec 14;50(6):1701134. doi: 10.1183/13993003.01134-2017. Print 2017 Dec. PMID 29242259
- [Result] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Result] Divo M, Cote C, de Torres JP, Casanova C, Marin JM, Pinto-Plata V, Zulueta J, Cabrera C, Zagaceta J, Hunninghake G, Celli B; BODE Collaborative Group. Comorbidities and risk of mortality in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 Jul 15;186(2):155-61. doi: 10.1164/rccm.201201-0034OC. Epub 2012 May 3. PMID 22561964
- [Result] Herrero MJ, Blanch J, Peri JM, De Pablo J, Pintor L, Bulbena A. A validation study of the hospital anxiety and depression scale (HADS) in a Spanish population. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):277-83. doi: 10.1016/s0163-8343(03)00043-4. PMID 12850660
- [Result] Ruiz Comellas A, Pera G, Baena Diez JM, Mundet Tuduri X, Alzamora Sas T, Elosua R, Toran Monserrat P, Heras A, Fores Raurell R, Fuste Gamisans M, Fabrega Camprubi M. [Validation of a Spanish Short Version of the Minnesota Leisure Time Physical Activity Questionnaire (VREM)]. Rev Esp Salud Publica. 2012 Oct;86(5):495-508. doi: 10.4321/S1135-57272012000500004. Spanish. PMID 23223762
- [Result] Guigoz Y, Lauque S, Vellas BJ. Identifying the elderly at risk for malnutrition. The Mini Nutritional Assessment. Clin Geriatr Med. 2002 Nov;18(4):737-57. doi: 10.1016/s0749-0690(02)00059-9. PMID 12608501
- [Result] Plaza V, Fernandez-Rodriguez C, Melero C, Cosio BG, Entrenas LM, de Llano LP, Gutierrez-Pereyra F, Tarragona E, Palomino R, Lopez-Vina A; TAI Study Group. Validation of the 'Test of the Adherence to Inhalers' (TAI) for Asthma and COPD Patients. J Aerosol Med Pulm Drug Deliv. 2016 Apr;29(2):142-52. doi: 10.1089/jamp.2015.1212. Epub 2015 Jul 31. PMID 26230150